CLINICAL TRIAL: NCT05082064
Title: Impact of Serum Bicarbonate and Electrolytes on Adverse Outcomes in Decompensated Cirrhotic Patients in Sohag University Hospital
Brief Title: Observational Prospective Study.at the End of the Study the Patients Will be Classified According to PH,Serum Bicarbonate and Serum Sodium Into 6 Groups and Statistical Analysis Will be Performed Using Spss
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Heba Allah Fadel Abdel Rahman, doctor,principle investigator, Sohag University
Other Study IDs: liver cirrhosis
Record Dates: First submitted 2021-09-10; First posted 2021-10-18 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- MELD score group A: MELD score :group A<25
  Interventions: Diagnostic Test: arterial blood gases and serum electrolytes
- MELD group B: Group B>25
  Interventions: Diagnostic Test: arterial blood gases and serum electrolytes
- MELD-PACO2 Group C: Group C<25
  Interventions: Diagnostic Test: arterial blood gases and serum electrolytes
- MELD -PACO2 Group D: Group D>25
  Interventions: Diagnostic Test: arterial blood gases and serum electrolytes
- MELD-BICARBONATE score Group E: Group E<23
  Interventions: Diagnostic Test: arterial blood gases and serum electrolytes
- MELD-BICARBONATE Group F: Group F>23
  Interventions: Diagnostic Test: arterial blood gases and serum electrolytes

INTERVENTIONS:
Diagnostic Test: arterial blood gases and serum electrolytes — arterial bloog gases parameters serum potassium serum sodium serum calcium

SUMMARY:
1-to identify the prognostic value of serum bicarbonate and serum electrolytes at time of admission and their association with development of complications ,length of hospital stay ,prognosis and mortality in hospitalized cirrhotic patient

DETAILED DESCRIPTION:
the purpose of this study will be explore the impact of data obtained for the arterial blood gas parameters and serum bicarbonate and electrolytes at the time of hospital admission on adverse clinical outcomes ,duration of length of hospital stay and mortality in patients with cirrhosis .Furthermore incorporation these parameters into model of end stage liver disease could help to improve the prognostic value of MELDscore in comparison to the prognostic value of traditional equation of original MELD and child score

ELIGIBILITY:
Inclusion Criteria:

patients with confirmed diagnosis of cirrhosis (age >18 years ) who will be admitted to internal medicine department or will be admitted to intermediate care unit

* willing and agree to be included in the study

Exclusion Criteria:

* patients without evidence of cirrhosis
* cirrhotic patients whom -younger than 18 years old

  * have diabetic ketoacidosis
  * with acute coronary syndrome
  * with fulminant liver failure
  * with heart failure
  * with organ transplantation
  * when arterial blood gases not be available
  * patient refusal
  * patient with HCC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the study protocol will be approved by ethical committee of sohag university of medicine written informed consent will be obtained from all participants
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-01-07 (Actual)

PRIMARY OUTCOMES:
will be ICU admitted | from the day of admission to the day of discharge from hospital or death during hospitalization
  will be admitted to ICU due to progression of the disease
  complications as shok,hepatorenal syndrome,severe infection,starting renal replacement therapy and icu intervention as mechanical ventilation using MELD score and child score depending on ABGparameters and serum electrolytes .

CONTACTS AND LOCATIONS:
Overall Officials: Heba allah Fadel, Doctor, Principal Investigator — Clinical trial organization
Locations (1):
- Heba Allah fadel abd elrahman, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Scheiner B, Lindner G, Reiberger T, Schneeweiss B, Trauner M, Zauner C, Funk GC. Acid-base disorders in liver disease. J Hepatol. 2017 Nov;67(5):1062-1073. doi: 10.1016/j.jhep.2017.06.023. Epub 2017 Jul 3. PMID 28684104